CLINICAL TRIAL: NCT02956447
Title: Administration of Kisspeptin in Patients With Hyperprolactinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002281; FD-R-5712 (Other Grant/Funding Number: FDA Office of Orphan Products Development)
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Results first posted 2024-08-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Hyperprolactinemia; Hypogonadism
Keywords: Kisspeptin; Hyperprolactinemia; GnRH; Hypogonadism
MeSH Terms: conditions — Hyperprolactinemia; Hypogonadism | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous Kisspeptin (Experimental): Blood sampling every 10 minutes over two 12-hour periods. One 12-hour period without any intervention. One 12-hour period consisting of administration of 10 boluses of kisspeptin 112-121 intravenously (IV).
  Interventions: Drug: Kisspeptin 112-121; Drug: GnRH
- Subcutaneous Kisspeptin (Experimental): Subcutaneous (SC) administration of kisspeptin 112-121 every 90 minutes over eight days.
  Interventions: Drug: Kisspeptin 112-121

INTERVENTIONS:
Drug: Kisspeptin 112-121 — 0.313 ug/kg - 2 ug/kg IV or SC
  Other Names: Metastin 45-54
Drug: GnRH — 0.075 ug/kg IV
  Other Names: gonadotropin-releasing hormone
  Arms: Intravenous Kisspeptin

SUMMARY:
The goal of this study is to learn more about how kisspeptin, a naturally occurring hormone, affects women with high levels of prolactin (also called hyperprolactinemia). Subjects in one group will undergo blood sampling every 10 minutes over two 12-hour periods (one 12-hour period without any intervention and one 12-hour period with intravenous (IV) kisspeptin administration). Subjects in the second group will receive subcutaneous (SC) kisspeptin every 90 minutes for eight days.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* confirmed diagnosis of elevated levels of prolactin measured via blood test,
* no pituitary adenoma OR a microprolactinoma (<10 mm). Patients with a macroprolactinoma confirmed on MRI imaging will be excluded,
* no history of a medication reaction requiring emergency medical care,
* no illicit drug use or excessive alcohol consumption (>10 drinks/week),
* not currently seeking fertility, breastfeeding or pregnant,
* no history of bilateral oophorectomy,
* willing to complete a dopamine agonist washout and/or oral contraceptive washout,
* normal physical exam and laboratory studies within protocol reference range.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
After primary results are published, the authors will provide individual participant data upon request as long as it does not conflict with state or institutional regulations

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Kisspeptin | Subcutaneous Kisspeptin
Started | 21 | 15
Completed | 10 | 5
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Kisspeptin | Subcutaneous Kisspeptin | Total
Number analyzed (Participants) | 21 | 15 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 15 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (8.3) | 30.4 (8.4) | 29.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 2 | 11
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 9 | 7 | 16
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 21 | 15 | 36

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Number of Luteinizing Hormone (LH) Pulses Over 10 Hours
Description: Average change in LH pulse frequency at baseline and during kisspeptin IV administration
Time Frame: Up to 14 days
Population: No analysis of this outcome was performed for the Subcutaneous Kisspeptin Arm. These individuals did not undergo IV kisspeptin delivery.
Measure: Mean (Standard Deviation); unit: pulses per 10 hour period
Arm/Group | Intravenous Kisspeptin | Subcutaneous Kisspeptin
Number analyzed (Participants) | 11 | 0
pulses per 10 hour period | 3.000 (3.066) |

2. Primary Outcome: Number of Participants With Evidence of Follicle Growth From Subcutaneous Kisspeptin
Description: Ultrasound evidence of increased follicle size over the course of SC kisspeptin administration
Time Frame: Evaluated over eight days
Population: No analysis of this outcome was performed for the Intravenous Kisspeptin Arm. These individuals did not undergo SC kisspeptin delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Subcutaneous Kisspeptin | Intravenous Kisspeptin
Number analyzed (Participants) | 5 | 0
Participants | 3 |

3. Secondary Outcome: Average Change in LH Pulse Amplitude
Description: Average change in LH pulse amplitude at baseline and during IV kisspeptin administration
Time Frame: Up to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Intravenous Kisspeptin | Subcutaneous Kisspeptin
Number analyzed (Participants) | 11 | 0
mIU/mL | -0.5764 (8.061) |

ADVERSE EVENTS:
Time Frame: From the time of documented informed consent until completion of study procedures (an average of 3 months).
Arm/Group | Intravenous Kisspeptin | Subcutaneous Kisspeptin
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/15
Other Adverse Events (participants affected / at risk) | 10/21 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Kisspeptin (N=21) | Subcutaneous Kisspeptin (N=15)
Headache (Nervous system disorders) | 5 (6) | 2 (5)
Fatigue (General disorders) | 2 (2) | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT02956447/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT02956447/ICF_001.pdf